CLINICAL TRIAL: NCT03045692
Title: Reliable Methods to Assess Kidney Function for Drug Dosage Adjustments in Critically Ill Patients - Comparison of Timed Clearance of Creatinine and Creatinine Based Estimated GFR
Brief Title: Assessment of Kidney Function for Drug Dosage Adjustments in Critically Ill Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jung Eun Lee, Associate professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2016-12-147-003
Record Dates: First submitted 2017-02-05; First posted 2017-02-07 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: ICU Patients
Keywords: drug dosing, eGFR, CCr

STUDY DESIGN:
Intervention Model Description: Double blind randomized trial
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): creatinine based eGFR (which is not revised value with standardized body surface area, that is, 1.73m2) are used to decide colistin maintenance dosage.
  Interventions: Diagnostic Test: kidney function assessment by creatinine based eGFR
- Study group (Experimental): 4 hour creatinine clearance is used to decide colistin maintenance dosage.
  Interventions: Diagnostic Test: kidney function assessment by 4 hour creatinine clearance

INTERVENTIONS:
Diagnostic Test: kidney function assessment by 4 hour creatinine clearance — 4 hour creatinine clearance is used to decide colistin maintenance dosage.
  Arms: Study group
Diagnostic Test: kidney function assessment by creatinine based eGFR — creatinine based eGFR (which is not revised value with standardized body surface area, that is, 1.73m2) are used to decide colistin maintenance dosage.
  Arms: Control group

SUMMARY:
The aim of the study is to determine if colistin dosage adjustment using 4hr CrCl contribute to better clinical outcomes compared with drug dosage adjustment using eGFR in critical ill patients. In control group, colistin maintenance dosage will be decided using serum creatinine based eGFR (in ml/min). In study group, colistin maintenance dosage will be decided using 4hr CrCl.

DETAILED DESCRIPTION:
1. Screening periods (From 'informed consents' to 'randomization')

   * Check of inclusion/exclusion criteria ② Measurement of 4hr CrCl & eGFR in ml/min

     * calculation of maintenance dose ③ Baseline characteristics & laboratory findings ④ Randomization
2. Colistin dosage Loading dose : 5 x body weight (not exceeding 300mg) Maintenance dose (after 12 hours from loading dose)

   : 2.5 x ([1.5 x GFR] + 30) (divided doses every 12hours), GFR in ml/min

   During the study period, daily morning serm creatinine levels are measured. Whenever serum creatinine concentration changes by more than 10% compared with baseline, 4hr CrCl will be mearued. At the every time of 4hr CrCl measurements, colistin dose wil be modified according to new GFR values (4hr CrCl in study group, eGFR in control group)
3. Blood sampling for Colistin trough level measurement Peripheral blood will be sampled twice between 72 hrs and 144 hours after loading dose, just before colistin infusion. The samples were collected in heparined tubes and centrifuged at 4 °C within 1 hr of collection. The resulting plasma was stored at - 70°C . And two values will be averaged out.
4. End of randomization (7 days after colistin initiation) ① Nephrotoxicity ② Treatment outcome microbiological outcome: eradication / no eradication clinical outcome: complete response / partial response / treatment failure

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged over 18
2. Patients in intensive care unit received colistin for the microbiologically documented cases associated with carbapenem-resistant gram negative bacilli.

Exclusion Criteria:

1. Patients who received colistin empirically.
2. Patients who received renal replacement therapy due to acute kidney injury or end-stage renal disease
3. Patients whose urine output was less than 0.5cc/kg/hr for 6 hrs
4. Patients who underwent hematopoietic stem cell transplantation
5. Patients who disagree with this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Estimated)
Dates: Start 2017-02-13 (Estimated); Primary Completion 2019-02-28 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
composite outcome (combination of nephrotoxicity or treatment failure) | 7 days after colistin initiation
  Nephrotoxicity means development of AKI (according to RIFLE criterior) Treatment failure menas clinically 'no response'

SECONDARY OUTCOMES:
colistin trough level, renal clearance of colistin | 7 days after colistin initiation
ICU stay duration | till discharge (Max. 3 months)
Total duration of colistin treatment | till discharge (Max. 3 months)
Need for renal replacement therapy | 7 days after colistin initiation
In-ICU mortality (infection-attributed mortality) | till discharge (Max. 3 months)

IPD SHARING:
Plan to Share IPD: No